CLINICAL TRIAL: NCT06024304
Title: Does an Integrated Dual Screw Design Improve Biomechanics and Function Following Fixation of Unstable Intertrochanteric Femur Fractures: a Randomized Pilot Trial (InterTAN)
Brief Title: InterTAN: Integrated Dual Screw Design Improve Biomechanics/Function Following Fixation Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul E. Matuszewski (Other)
Responsible Party: Sponsor-Investigator, Paul E. Matuszewski, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO-22-INTERTAN
Record Dates: First submitted 2022-04-13; First posted 2023-09-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Fracture of Hip
Keywords: Surgical Fixation; Cephalomedullary nail
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Pilot, patient blinded randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trigen InterTan (Active Comparator): Patients in this arm will be implanted with the cephalomedullary nail Trigen InterTan manufactured by Smith & Nephew.
  Interventions: Device: Trigen InterTAN
- Synthes TFNA (Active Comparator): Patients in this arm will be implanted with the single-screw device TFNA manufactured by DePuy Synthes.
  Interventions: Device: Synthes TFNA

INTERVENTIONS:
Device: Synthes TFNA — Surgical fixation with single-screw device Synthes TFNA; Pelvic fractures will be repaired utilizing single-screw device Synthes TFNA.
  Arms: Synthes TFNA
Device: Trigen InterTAN — Surgical fixation with Smith and Nephew Trigen InterTAN cephalomedullary long nail; Pelvic fractures will be repaired utilizing Smith and Nephew Trigen InterTAN.
  Arms: Trigen InterTan

SUMMARY:
The goal of this pilot, patient blinded randomized trial is to develop a mechanistic understanding of gait following fixation of unstable intertrochanteric hip fractures and return to function and pain control. The guiding hypothesis that will be tested in a subsequent clinical trial is that the InterTAN when compared to standard lag-screw cephalomedullary nails will have decreased post operative pain, earlier return to symmetric weight bearing, and quicker return to pre-injury functioning levels.

DETAILED DESCRIPTION:
Aim 1: Determine the feasibility of conducting a randomized trial assessing gait mechanics as well as outcomes following unstable intertrochanteric femur fractures treated with cephalomedullary nails. This will be achieved by performing a pilot randomized trial comparing the InterTAN versus a single-screw design cephalomedullary nail (SSCMN). Deliverable: Preliminary data to support a larger randomized trial powered on either mechanical assessments or patient reported outcomes. Feasibility of conducting comprehensive biomechanical and patient related outcome measurements in the geriatric hip fracture population.

Aim 2: Determine the pathway to return to function and symmetric weight bearing. Load bearing will be assessed through insole monitoring during their inpatient stay and 2-weeks post-op. Additionally, analysis will be performed to measure gait for hip motion, loading, strength and functional assessments at 6,12, and 26 weeks post-op. Patients will also be assessed at 1-year for reported function as well. Hypothesis: Patients in the InterTAN group will have faster return to symmetrical weight bearing/motion and earlier return to function. Deliverable: Longitudinal data assessing return to function and weight bearing in intertrochanteric femur fractures.

Aim 3: Determine if use of the InterTAN device when compared to SSCMN results in decreased pain following unstable intertrochanteric femur fractures. Patients will be enrolled in a prospective trial with standardized pain control regimen, assessing patients for pain during their hospital stay using Area Under the Curve Analysis of Visual Analogue Pain Scores at 24, 48 and 72 hours. Similarly, opioid usage in morphine milligram equivalents will be assessed. Pain will be assessed at follow-up visits 6, 12, 26, 52 weeks. Hypothesis: The InterTAN will result in decreased pain in the immediate post-operative period and in sub-acute post-operative period.

Aim 4: Determine if the use of the InterTAN device when compared to SSCMN results in decreased healthcare utilization. Participation with therapy, hospital length of stay, discharge disposition, and time-spent in rehabilitation facility will be assessed. Hypothesis: Patients in the InterTAN group will be more likely to be discharged home, participate with therapy more, have decreased length of stay in both inpatient and outpatient units. Deliverable: Data to inform the power analysis for a larger prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Non-pathologic fractures
* OTA/AO classification 31A2, 31A3 fractures
* Ability to participate in 4-MET equivalent activities without ambulatory assistance prior to injury

Exclusion Criteria:

* Inability to consent
* Inability to participate in follow-up activities
* History of chronic pain / current opioid treatment
* Pre-injury ambulatory status requiring assistance device
* Neurological condition altering gait or sensation (e.g. History of stroke with altered gait, peripheral neuropathy).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported physical function | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function Questionnaire is a 53 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates less physical function.
Change in self-reported pain | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Questionnaire is a 56 question survey with a five point Likert scale ranging from 1 to 5 where a higher number indicates increased interference due to pain.

SECONDARY OUTCOMES:
Change in Functional Independence Measure | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  The Functional Independence Measure (FIM) is a tool used to measure the level of disability as well as the change in patient status. FI is comprised of 18 items, grouped into 2 subscales - motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.
Change in pain assessment | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  Brief Pain Inventory (BPI) will be used to measure pain intensity. This is a four-item scale that measures current, worst, least, and average pain. Each of these four items are measured on a numeric scale from 0 to 10 with 0 being ''no pain'' and 10 being ''severe pain.''
Change in weight bearing | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  The ground reaction forces of the injured and non injured limb will be evaluated over the course of recovery to assess when loading between limbs becomes symmetric during their physical therapy.
Change in Visual Analog Pain Score | 2 weeks, 6 weeks, 12 weeks, 26 weeks, 12 months
  The visual analog pain score is a horizontal line with a scale ranging from 0 to 10 where a higher number indicates more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Matuszewski, MD, Principal Investigator — University of Kentucky

IPD SHARING:
Plan to Share IPD: No